CLINICAL TRIAL: NCT00000865
Title: A Phase I Safety and Pharmacokinetic Study of 1592U89 Alone and In Combination With Other Antiretroviral Agents in Infants and Children With HIV Infection
Brief Title: The Safety and Effects of 1592U89 Used Alone or in Combination With Other Anti-HIV Drugs in HIV-Infected Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 330; 11302 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To assess the steady state pharmacokinetic features, tolerance, and safety of orally administered 1592U89, given alone or in combination with other antiretroviral medications, in HIV infected infants and children. To establish doses of 1592U89 appropriate for future pediatric Phase II/III clinical trials.

On the basis of the preclinical and clinical studies, 1592U89 appears to be a promising agent for treatment of HIV infection in children, either as an alternative to currently employed agents, or in combination therapy regimens. A liquid formulation of the drug is available; thus concurrent development of 1592U89 for children and adults is possible.

DETAILED DESCRIPTION:
On the basis of the preclinical and clinical studies, 1592U89 appears to be a promising agent for treatment of HIV infection in children, either as an alternative to currently employed agents, or in combination therapy regimens. A liquid formulation of the drug is available; thus concurrent development of 1592U89 for children and adults is possible.

In part 1, patients will receive 1592U89 monotherapy for 12 weeks. Patients will be assigned initially to a low dose of 1592U89 (Dose A). Those patients who tolerate the drug for at least six weeks without a toxicity of grade 3 or above attributable to study drug will have their 1592U89 dose increased (Dose B). If none of those patients experience a life threatening event attributable to study drug, subsequent enrollees will be assigned initially to Dose B. In part 2, each participant will be assigned randomly (1:1:1:1) within their age and Part 1 regimen stratum to one of the four agents: Zidovudine (ZDV), Stavudine (d4T), Didanosine (ddI) or Lamivudine (3TC) in combination with 1592U89.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* IVIG.
* Erythropoietin, granulocyte colony stimulating factor and granulocyte macrophage colony stimulating factor (for management of hematologic toxicity).

Patients must have:

* Documented HIV-1 infection.
* Laboratory evidence of immunosuppression or symptomatic HIV disease.
* Parent or legal guardian able and willing to provide signed informed consent.

Prior Medication: Required:

* HIV infected infants and children will be eligible for the trial if they have received greater than 56 days of previous antiretroviral therapy.

NOTE:

* Those children who participated in the single dose phase I study of 1592U89 and satisfy all other criteria for inclusion may have received <= 56 days of previous antiretroviral therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Grade 3 or greater abnormalities in any toxicity monitoring laboratory tests at baseline.
* Presence of an acute opportunistic infection requiring therapy at the time of enrollment.
* Intractable or chronic diarrhea or vomiting.

Concurrent Medication:

Excluded:

* Chemotherapy for active malignancy.
* Concurrent use of antiretroviral agents other than those provided by the study, biologic response modifiers, human growth hormone, systemic corticosteroids (>= 14 days duration), probenecid, I.V. pentamidine, immunomodulators (other than intravenous immunoglobulin), or other investigational drugs.

Patients with any of the following prior conditions or symptoms are excluded:

- History of intolerance to any of the study drugs.

Ages: 3 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32
Dates: Study Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kline M, Study Chair; Van Dyke R, Study Chair; Yogev R, Study Chair; Shenep J, Study Chair
Locations (7):
- United States (7):
  - Usc La Nichd Crs, Los Angeles, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas

REFERENCES:
- [Background] Hughes W, McDowell J, L Adams, Flynn P, Hetherington S, Kline M, Shenep J, Yogev R, Lafon S. Evaluation of the novel nucleoside 1592U89 in a phase I safety and pharmacokinetics (PK) study in HIV-infected infants and children. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:115